CLINICAL TRIAL: NCT00810875
Title: Analysis of the Maternal-fetal Interface During Maternal Hepatitis C Virus Infection and Influenza Virus Vaccination
Brief Title: Study of Maternal Hepatitis C Infection and Influenza Vaccination in Pregnancy
Status: Terminated | Type: Observational
Why Stopped: Terminated due to lack of enrollment
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: HCVP-1
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Hepatitis C
Keywords: pregnancy; immunity; cord blood; influenza vaccines; disease transmission, vertical
MeSH Terms: conditions — Hepatitis C; Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, peripheral and cord blood mononuclear cells, placental tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- hepatitis C: pregnant women with hepatitis C virus infection and their infants
- controls: pregnant women without hepatitis C infection and their infants

SUMMARY:
The purpose of this study is to determine if hepatitis C virus and influenza virus vaccine components can cross the placenta and stimulate an immune response in the fetus.

DETAILED DESCRIPTION:
The rate of mother-to-child transmission of hepatitis C virus (HCV) is only 5%, even though the level of fetal exposure to the virus during pregnancy is probably much higher. How can the fetus avoid infection in so many cases? We believe the fetal immune system is not immature as has previously been thought, but instead plays an active role in protecting the fetus from infection. In this study, we aim to better understand the immune response of the fetus against maternal HCV infection. In addition, since the fetus has been shown in some cases to make an immune response against vaccines given to the mother during pregnancy, we also aim to study the fetal immune response against maternal influenza virus vaccination. We plan to study 50 HCV-positive pregnant women and their infants (study group) and compare them to 20 HCV-negative pregnant women and their infants (control group). We estimate that approximately 30 women in the study group will have received the influenza virus vaccine. We will analyze 3 important components of mother-to-child transmission: (1) the maternal immune response against HCV and influenza virus vaccine during and after pregnancy; (2) the baby's immune response to these agents at birth, 9-15 months, and 24 months; and (3) the placenta, for the presence of HCV particles or influenza virus vaccine components. The results of this study may have implications for the prevention of mother-to-child transmission of HCV and other infections, as well as for the development of novel vaccination strategies.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women 18 years of age or older
* infants born to these women from this pregnancy
* hepatitis C virus antibody and RNA positive (for study group)
* hepatitis C virus antibody and RNA negative (for control group)

Exclusion Criteria:

* HIV infection
* hepatitis B infection
* plan to use cord blood for another purpose

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both groups will be selected from an outpatient obstetrics clinic.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Detection and characterization of cord blood immune responses against hepatitis C virus and influenza virus vaccine | single time point (birth)

SECONDARY OUTCOMES:
Characterization of immune responses in infants against hepatitis C virus and influenza virus vaccine | 2 time points (9-15 months and 24 months)
Detection and characterization of immune responses against hepatitis C virus and influenza virus vaccine in mothers | 2 time points (prenatal and postpartum time points)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M McCune, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, University of California, San Francisco, San Francisco, California, United States